CLINICAL TRIAL: NCT04853602
Title: IFx-Hu2.0 Expanded Access Program
Status: Available | Type: Expanded Access
Sponsor: TuHURA Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IFx-Hu2.0 Expanded Access
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cutaneous Melanoma, Stage III; Cutaneous Melanoma, Stage IV; Merkel Cell Carcinoma; Cutaneous Squamous Cell Carcinoma
Keywords: CM; MCC; cSCC; pDNA; plasmid DNA; pAc/emm55; IFx-Hu.20; Immunotherapy; Gene Therapy; Immunology; Oncology; Immuno-Oncology
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Biological: IFx-Hu2.0 — The investigational drug product IFx-Hu2.0 is composed of the drug substance pAc/emm55 (pDNA) complexed with the two excipients in vivo-jetPEI® (linear polyethylenimine), a transfection reagent, and dextrose, a pDNA/polyethylenimine complex stabilizer.
  Therapeutic Classification:
  * Immunomodulatory Agent
  Route of Administration:
  * Intralesional (i.e. injection of cutaneous, subcutaneous or nodal lesions)
  Mechanism of Action:
  * Injection of IFx-Hu2.0 into the lesion facilitates the expression of the immunogenic Emm55 protein by the tumor cells.
  Physiological Effect:
  * Expression of the emm55 gene by the tumor cells triggers immune recognition of tumor-specific and -associated antigens which leads to innate and adaptive immune responses. In addition to priming anti-tumor immunity in immune checkpoint inhibitor (ICI)-naïve patients, this could re-sensitize patients with primary or secondary ICI clinical resistance.
  Other Names: pAc/emm55

SUMMARY:
Expanded access requests for IFx-Hu2.0 may be considered for the treatment of adult patients (greater than or equal to 18 years of age) with stage III through IV cutaneous melanoma, advanced Merkel cell carcinoma (MCC), or advanced cutaneous squamous cell carcinoma (cSCC) who have failed all available treatment options.

To request access, use Responsible Party contact information provided in this record..

ELIGIBILITY:
Inclusion Criteria:

* To request more information use Responsible Party contact information provided in this record

Exclusion Criteria:

* To request more information use Responsible Party contact information provided in this record

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Bunch BL, Kodumudi KN, Scott E, Morse J, Weber AM, Berglund AE, Pilon-Thomas S, Markowitz J. Anti-tumor efficacy of plasmid encoding emm55 in a murine melanoma model. Cancer Immunol Immunother. 2020 Dec;69(12):2465-2476. doi: 10.1007/s00262-020-02634-4. Epub 2020 Jun 18. PMID 32556443